CLINICAL TRIAL: NCT00756769
Title: Systemic Lupus Erythematosus in Gullah Health
Acronym: SLEIGH
Status: Recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: MUSC HR10852; P60AR049459 (NIH)
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: African Americans
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients with SLE
- 2: Related unaffected controls
- 3: Unrelated unaffected controls

SUMMARY:
Systemic lupus erythematosus (SLE) is an autoimmune disease characterized by the production of autoantibodies, multiple organ involvement, and diverse clinical symptoms and immunologic manifestations. African Americans are at a disproportionately higher risk of developing SLE, develop SLE at an earlier age, and have increased morbidity and mortality compared with European Americans. Our central study hypothesis is that there are specific genetic factors that interact with environmental exposures leading to the development of SLE. The African American Gullah population from the Sea Islands of South Carolina and Georgia are unique in their genetic homogeneity with minimal non-African genetic admixture, making them an ideal cohort to address questions of environmental and genetic influence on the development and progression of SLE.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 years and above;
* Self-identified as African-American "Gullah" from the Sea Island region of South Carolina;
* Have had at least 4 of the 11 diagnostic criteria for SLE as designated by the American College of Rheumatology (ACR), be a relative of a known SLE patient, or be an unrelated healthy Gullah control;
* Ability to speak and understand English;
* Ability and willingness to give informed consent

Exclusion Criteria:

* Race defined by participant as other than Black or African-American;
* Being a prisoner, mentally ill patient, or institutionalized individual;
* Unwilling or unable to give informed consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sea Island Community
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2003-04; Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Diane L. Kamen, MD, MSCR, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Kamen DL, Barron M, Parker TM, Shaftman SR, Bruner GR, Aberle T, James JA, Scofield RH, Harley JB, Gilkeson GS. Autoantibody prevalence and lupus characteristics in a unique African American population. Arthritis Rheum. 2008 May;58(5):1237-47. doi: 10.1002/art.23416. PMID 18438839